CLINICAL TRIAL: NCT06104592
Title: Phase 2, Single-Arm Trial of Comprehensive Ablative Bridging Irradiation (CABI) Prior to CD19 CAR-T Cell Therapy in High-Risk, Relapsed or Refractory Large B Cell Lymphoma in Patients With Bulky Disease
Brief Title: Single-Arm Comprehensive Ablative Bridging Irradiation I Prior to CD19 CAR-T In High-Risk R/R LBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22113
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma; Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy and CAR T-Cell Infusion (Experimental): Following T-cell apheresis for CD19 CAR T-cell therapy, eligible enrolled study participants patients will undergo Comprehensive Ablative Bridging Irradiation (CABI) to all pretreatments lesions that are able to be feasibly and safely treated by the treating radiation oncologist. Upon completion of bridging radiotherapy, patients will undergo lymphodepleting chemotherapy period (Days -5, -4, -3) followed by axi-cel infusion (Day 0).
  Interventions: Radiation: Comprehensive Ablative Bridging Irradiation (CABI); Biological: Chimeric Antigen Receptor T-Cell Therapy

INTERVENTIONS:
Radiation: Comprehensive Ablative Bridging Irradiation (CABI) — Participants will receive radiation therapy to all pretreatment lesions that are able to be feasibly and safely treated.
Biological: Chimeric Antigen Receptor T-Cell Therapy — Yascarta is an autologous anti-CD19 CAR T cell therapy manufactured from the patient's own T cells, which have been extracted and then reprogrammed with CAR molecules to help the T cells recognize cancer cells. The reengineered T cells are infused back into the patient to attack the cancer.
  Other Names: Axi-Cel; Yascarta

SUMMARY:
This is a phase 2, single-arm, open-label study to evaluate the safety and efficacy of comprehensive bridging radiation therapy prior to CD19 CAR T-cell therapy for large B-cell lymphoma patients with bulky disease, defined as any lesion ≥5 cm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) who plan to receive treatment at the Moffitt Cancer Center will be eligible.
* Must have ability to comprehend and the willingness to sign written informed consent for study participation.
* Eligible to receive CAR T-cell therapy (axicabtagene ciloleucel) for LBCL and histological variants approved by the standard of care label
* ECOG performance status 0 to 2.
* At least one high-risk lesion, defined as measuring ≥ 5 cm, that is targetable for radiotherapy per investigator assessment.
* Ability to undergo comprehensive bridging radiation, defined as radiation to all visible sites of disease.
* No evidence or suspicion of active central nervous system (CNS) involvement of lymphoma
* Adequate bone marrow and organ function as defined in protocol.

The effects of therapeutic agents used in this trial on developing human fetus are unknown, and because of this, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation as outlined in criteria below:

* Men must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow up and must refrain from donating sperm during this period. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants in their understanding confirmed.
* Women of childbearing potential must have a negative serum or urine pregnancy test at screening and at time of radiation treatment planning, per standard of care and departmental standard operating procedure. Patients must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
* Women of non-childbearing potential (i.e., surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥12 months of amenorrhea) are eligible.

Exclusion Criteria:

* Patients who are currently receiving or who have received any other investigational study agent ≤4 weeks prior to screening visit are ineligible
* Prior treatment with chimeric antigen receptor (CAR) T-cell therapy
* Inability to safely deliver comprehensive radiation therapy to all sites of disease per treating radiation oncologists' discretion
* Participants with clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from screening, New York Health Association III or IV heart failure, and circulatory collapse requiring vasopressor or inotropic support.
* Participants with arrhythmias that are not stable on a medical management program within 2 weeks of screening are also excluded.
* Evidence of active uncontrolled/untreated infection (viral, bacterial, fungal, opportunistic) of any origin.
* Known positive Human immunodeficiency virus (HIV) status.
* Participants with evidence of active and/or chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection, HCV must have a negative nucleic acid test post-treatment or spontaneous clearance.
* Participants who require the concurrent use of chronic systemic steroids or immunosuppressant medications. Steroids should not be given within 5 days prior to leukapheresis. Concomitant bridging steroids (Section 6.6) are allowed after leukapheresis.
* Any condition that would, in the investigator's judgement, interfere with full participation in the study and attending required study visits (if outpatient); pose a significant risk to the participant; or interfere with interpretation of study data.
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation including ability to safely undergo radiation treatment planning and delivery.
* Women of childbearing potential who are pregnant or breastfeeding. Females who have undergone surgical sterilization or who have been postmenopausal for at least 12 months are not considered to be of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | at 12 months
  PFS will be measured by date of CAR T-cell infusion until first occurrence of in-field, local, or distant progression, or death. If none of these events occur, patients will be censored on date of last contact.

SECONDARY OUTCOMES:
Rate of local relapse (i.e., relapse of lymphoma at a body site that received bridging radiation therapy) | up to 12 months
  Rate of local relapse determined by evidence of disease at a body site that received bridging radiation therapy.
Rate of distant relapse (i.e., relapse of lymphoma at a body site that did not receive bridging radiation therapy) | up to 12 months
  Rate of distant relapse determined by evidence of disease at a body site that did not receive bridging radiation therapy.
Number of serious adverse events attributed to bridging radiotherapy | Up to 12 months
  Number of serious adverse events that can be attributed to bridging radiotherapy
Number of serious adverse events attributed to CAR T-cell infusion | Up to 12 months
  Number of serious adverse events that can be attributed to CAR T-cell infusion
Number of participants experiencing severe cytokine release syndrome (CRS) | at 30 days after CAR T infusion
  Number of participants experiencing severe CRS (grade 3 or higher by ASTCT criteria) in the first 30 days after CAR T-cell infusion.
Number of participants experiencing severe immune cell associated neurotoxicity syndrome (ICANS) | at 30 days after CAR T infusion
  Number of participants experiencing severe ICANS (grade 3 or higher by ASTCT criteria) in the first 30 days after CAR T-cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jain, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided